CLINICAL TRIAL: NCT01817010
Title: Strength and Function Following Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09-1121
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Total Hip Arthroplasty
Keywords: Total Hip Arthroplasty; Muscle Strength; Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — MCC protocol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multi-Component Rehabilitation (CMC) (Experimental): The CMC group will receive a multi-component program focused on rehabilitation of the abdominal and core musculature, neuromuscular re-education through therapeutic exercise as well as hip and knee muscle strengthening beginning 2 weeks after THA.
  Interventions: Behavioral: Multi-Component Rehabilitation (CMC)
- Control (CON) (Active Comparator): The CON group will participate in physical therapist recommended activities based on their home rehabilitation and then will complete the same CMC rehabilitation intervention beginning 10 weeks after THA.
  Interventions: Behavioral: Control (CON)

INTERVENTIONS:
Behavioral: Multi-Component Rehabilitation (CMC)
  Arms: Multi-Component Rehabilitation (CMC)
Behavioral: Control (CON)
  Arms: Control (CON)

SUMMARY:
To determine if patients who receive an 8 week, comprehensive, multi-component rehabilitation program (CMC) have better strength and functional performance compared to a control group (CON).

The investigators hypothesize that functional performance and strength in the muscles surrounding the hip and the knee will be greater in the multi-component rehabilitation group compared to the control group.

DETAILED DESCRIPTION:
The participants will be enrolled and following surgery, randomized into one of two treatment groups (CMC or CON). Prior to randomization, both groups will participate in two weeks of home rehabilitation consisting mobility training and activities of daily living. After randomization, the CMC group will receive physical therapy 2x/ week for 8 weeks from a licensed physical therapist and member of the investigative team starting 2 weeks after Total Hip Arthroplasty (THA). The CON group will continue activities provided by their home rehabilitation therapist for 8 weeks. The CON group will then participate in the CMC intervention beginning 10 weeks after THA. These patients will complete pre-operative and post-operative testing as described above.

The CMC group will receive a multi-component program focused on rehabilitation of the abdominal and core musculature, neuromuscular re-education through therapeutic exercise as well as hip and knee muscle strengthening beginning 2 weeks after THA. The CON group will participate in physical therapist recommended activities based on their home rehabilitation and then will complete the same multi-component rehabilitation intervention beginning 10 weeks after THA.

ELIGIBILITY:
Inclusion Criteria:

* receiving a total hip replacement secondary to MD diagnosed end-state osteoarthritis only
* cognitive status that allows patients to consistently comprehend and repeat back directions regarding the details of the study.

Exclusion Criteria:

* HbA1c levels greater than 7% based on medical records
* neurological, vascular or cardiac problems that limit function
* moderate or severe osteoarthritis or other orthopaedic conditions in the non-operated lower extremity
* lower back pain which interferes with activities of daily living
* diagnosed disease which affects muscle function (Parkinson's, Fibromyalgia, Multiple Sclerosis)
* history of vestibular dysfunction
* body mass index greater than 40
* alcoholism or drug abuse

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2012-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Stair Climbing Time | preoperatively and post operatively at 6, 10, 18 and 28 weeks
  Time to ascend and descend 12 stairs.

SECONDARY OUTCOMES:
Functional Performance Tests | preoperatively and post operatively at 6, 10, 18 and 28 weeks
  Health status and activity questionnaires (SF-36, WOMAC, UCLA score), timed up and go test, sit to stand performance, 6 minute walk test, timed Single Leg balance on variable surfaces, Fullerton Assessment of Balance and the modified Trendelenburg test
Isometric Muscle Strength | preoperatively and post operatively at 6, 10, 18 and 28 weeks
  Isometric strength of the hip flexors, extensors, abductors and knee extensors and flexors.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Stevens-Lapsley, PT,PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Anschutz Medical Campus, Aurora, Colorado, United States